CLINICAL TRIAL: NCT03771287
Title: Learning to Listen in Noise: A Double-blind Randomized Control Trial of a New Hearing Aid Noise Reduction System
Brief Title: Hearing Aid Noise Reduction in Pediatric Users (Oticon Study)
Acronym: OtiS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Oticon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-5953
Record Dates: First submitted 2018-11-27; First posted 2018-12-11 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-01

CONDITIONS: Hearing Impairment; Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded randomized control trial of OpenSound Navigator (OSN) enabled/disabled hearing aids. Only the fitting audiologist will know if the OSN algorithm is enabled or disabled in the research hearing aids. Will be un-blinded after data collection is complete in order to carry out group comparison analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OpenSound Navigator (OSN) Hearing Aid (Experimental): Participants will be fit with Oticon OPN™ behind-the-ear hearing aids with the OpenSound Navigator algorithm enabled. Participants are to use the hearing aids at least an average of 8 hours per day over the course of 6-8 months.
  Interventions: Device: Oticon OpenSound Navigator speech enhancement algorithm
- omni-directional Hearing Aid (Active Comparator): Participants will be fit with Oticon OPN™ behind-the-ear hearing aids with the Omni-directional microphone system enabled. Participants are to use the hearing aids at least an average of 8 hours per day over the course of 6-8 months.
  Interventions: Device: Oticon omni-directional microphone algorithm

INTERVENTIONS:
Device: Oticon OpenSound Navigator speech enhancement algorithm — OpenSound Navigator (OSN) is a speech enhancement algorithm developed by Oticon. The feature is built in Oticon's current OPN™ hearing aid platform and can be adjusted and disabled in the programming. It is designed to automatically enhance speech while reducing unwanted background noise to improve communication for the user.
  Other Names: OSN
  Arms: OpenSound Navigator (OSN) Hearing Aid
Device: Oticon omni-directional microphone algorithm — Omni-directional microphone setups come standard for all Oticon hearing aid models. The hearing microphones have equal sensitivity across all directions.
  Other Names: omni-directional mic
  Arms: omni-directional Hearing Aid

SUMMARY:
The purpose of this study is to evaluate the efficacy of OpenSound Navigator (OSN), a hearing aid speech-enhancement algorithm developed by Oticon, as treatment for pediatric hearing aid users. Using a double-blind experimental design, the investigators aim to compare two treatment groups of pediatric (ages 6-12) patients with symmetrical sensorineural hearing losses ranging from the mild to moderately-severe degree. One group will be fit with bilateral Oticon OPN™ behind-the-ear hearing aids set with an omni-directional microphone setting. The other group will be fit with the same hearing aid model with the OSN algorithm enabled. Participants from the groups will be age and audiogram-matched. The investigators will evaluate hearing aid benefit through word recognition in noise (behavioral testing) and everyday hearing/listening abilities (parental/legal guardian reported) at hearing aid fitting and 6-8 months post fitting.

DETAILED DESCRIPTION:
OpenSound Navigator (OSN) is a speech enhancement hearing aid algorithm developed by Oticon that utilizes an adaptive directional microphone system with an automatic gain control noise reduction program. This hearing aid feature is intended for adult hearing aid users and its potential benefits of speech, vocabulary and listening development in pediatric users has not been investigated. Here the investigators aim to evaluate the efficacy of OSN programming in pediatric hearing aid users (6-12 years of age) diagnosed with a symmetrical sensorineural hearing loss in the mild to moderately-severe range. The investigators will use a double-blind randomized control methodology of two participant matched (based on age and audiometric configuration) groups. The first group will include pediatric patients fit with bilateral Oticon OPN™ behind-the-ear hearing aids with the standard Omni-directional microphone setting enabled. Group two will include pediatric patients fit with the same hearing aid model with the OSN feature enabled. Participants will undergo standard audiometric diagnostic testing and will be fit with the hearing aids by a licensed clinical audiologist. Participants are required to wear the hearing aids full time (at least 8 hours per day average) during the duration of the study. The evaluation measures will include speech recognition testing in controlled background noise and the Speech, Spatial and Qualities of Hearing Scale questionnaire (completed by parents/legal guardian). Testing will be performed within a week of the hearing aid fitting and 6-8 months post fitting.

ELIGIBILITY:
Inclusion Criteria:

* children ages 6 to 13 years
* English as the primary home language
* positive for bilateral symmetrical mild to moderately-severe sensorineural hearing loss
* currently using hearing aids that were dispensed at least 18 months prior to enrollment of the study
* negative for major cognitive handicap or developmental delay that would prevent or restrict participation, as determined by the PI or designee
* negative for learning disability, for example attention-deficit/hyperactivity disorder, as determined by the PI or designee
* negative for serious neurological or psychiatric disease that would prevent or restrict participation, as determined by the PI or designee
* informed consent of parent/guardian
* assent of participating child if aged 11 years and over
* standard MRI inclusion criteria as set by the Cincinnati Children's Hospital Medical Center department of Radiology
* not currently pregnant or breast feeding
* willingness and ability of the participant and/or the participant's caregiver to comply with study requirements
* no history of medical neglect of caregiver

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Word Recognition Abilities at 6 to 8 Months | 6-8 months
  Aided speech perception in noise within a week of hearing aid fitting and again 6-8 months later.

SECONDARY OUTCOMES:
Change from Baseline Speech, Spatial Qualities of Hearing Scale (SSQ) Scores at 6 to 8 Months | 6-8 months
  Speech, Spatial and Qualities of Hearing Scale (SSQ), a survey utilizing an ordinal scale specifically measuring hearing aid benefit with regard to speech understanding, spatial awareness, perceptual quality of sound, and conversation, will be completed by parents/legal guardian within a week of the hearing aid fitting and after wearing the study hearing aids for 6-8 months. There are 4 survey sections. Section A: Speech has 8 questions, Section B: Spatial Hearing has 5 questions, Section C: Qualities of Hearing has 8 questions and Section D: Conversational Uses of Hearing has 5 questions. Each question uses a scale ranging from 0 (poorest possible outcome) to 100 (best possible outcome). Each section calculates an average score across the corresponding questions for a total of 4 individual scores.
Hearing aid use time | 6-8 months
  Average daily use of hearing aids.

CONTACTS AND LOCATIONS:
Overall Officials: David R Moore, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stewart HJ, Cash EK, Pinkl J, Nakeva von Mentzer C, Lin L, Hunter LL, Moore DR; CCHMC Division of Audiology. Adaptive Hearing Aid Benefit in Children With Mild/Moderate Hearing Loss: A Registered, Double-Blind, Randomized Clinical Trial. Ear Hear. 2022 Sep-Oct 01;43(5):1402-1415. doi: 10.1097/AUD.0000000000001230. Epub 2022 Jun 27. PMID 35758427